CLINICAL TRIAL: NCT01148238
Title: Autoimmune Diabetes: Disease Markers and Treatment of Latent Autoimmune Diabetes in Adults (LADA)
Brief Title: Autoimmune Diabetes: Markers of the Disease and Treatment of Latent Autoimmune Diabetes in Adults (LADA)
Status: Withdrawn | Type: Observational
Why Stopped: changed research plan
Sponsor: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Other Study IDs: AUTO
Record Dates: First submitted 2010-06-17; First posted 2010-06-22 (Estimated); Last update posted 2012-12-10 (Estimated); Status verified 2012-12

CONDITIONS: Autoimmune Diabetes
Keywords: Autoimmune diabetes; LADA; T-reg; cytokine
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Cytokines HLA T-reg
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Diabetes type 1 older than 10 years: Blood samples will be taken from 10 patients with diabetes type 1 older than 10 years and 10 healthy age-and sexmatched controls.
- Newly diagnosed type 1 diabetes: Blood samples will be taken from 10 patients with newly diagnosed type 1 diabetes and 10 healthy age-and sexmatched controls.
- LADA: Blood samples will be taken from 10 patients with LADA and 10 healthy age-and sexmatched controls.

SUMMARY:
Autoimmunity is the main cause of diabetes type 1 and an important factor as cause of Latent Autoimmune Diabetes in Adults (LADA). Recently, research has found that being deficient of T-reg cells is an important cause of autoimmunity. The study hypothesis are:

1. Patients with newly found diabetes type 1 have less T-reg than healthy.
2. Patients with newly found diabetes type 1 have less T-reg than patients with long duration of the illness.
3. The number of T-reg is negative associated with HLA-risk-haplotype.
4. The number of T-reg is negative associated with LADA.
5. Differences relating to inflammatory cytokines will be seen among patients with newly found diabetes type 1, but not among others.

DETAILED DESCRIPTION:
Research has worked out that b-cells are being destroyed by cytokines released from inflammatory cells. One hypothesis in that T-reg is a cause of autoimmunity, and that T-reg concentrations are low in patients with newly diagnosed diabetes type 1.

Blood samples will be taken from 10 patients with newly diagnosed type 1 diabetes, Latent Autoimmune Diabetes in Adults (LADA) and type 1 diabetes older than 10 years and the same amount of samples from healthy, age- and sex-matched blood donors. Markers of autoimmune diabetes will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* newly diagnosed diabetes type 1
* LADA
* diabetes type 1 older than 10 years

Exclusion Criteria:

* none

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 10 patients with newly diagnosed diabetes type 1. 10 healthy age- and sex matched blood donors.
  10 patients with LADA. 10 healthy age- and sex matched blood donors. 10 patients with diabetes type 1 older than 10 years. 10 healthy age- and sex matched blood donors.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2012-08; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
T-reg

SECONDARY OUTCOMES:
HLA, anti-GAD, anti-IA2, white blood count, CRP, fasting C-peptide, HbA1c

CONTACTS AND LOCATIONS:
Overall Officials: Valdemar Grill, M.D, PhD, Principal Investigator — Department of Cancer Research and Molecular Medicine